CLINICAL TRIAL: NCT02026817
Title: An Open-label, Randomized, Single-dose Crossover Study to Compare the Pharmacokinetics After the Administration of HCP1201 Tablet 750/10 mg and Coadministration of Metformin SR 750 mg and Rosuvastatin 10 mg in Healthy Volunteers
Brief Title: Comparison of PK After Administration of HCP1201 and Co-administration of Metformin SR 750mg and Rosuvastatin 10mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-MERO-104
Record Dates: First submitted 2014-01-01; First posted 2014-01-03 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCP1201 (Experimental): Participants received a single oral dose of the HCP1201 750/10 mg under fed condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: HCP1201 750/10mg
- Metformin and Rosuvastatin (Active Comparator): Participants received a single oral dose of coadministration of Metformin SR 750 mg and Rosuvastatin 10 mg under fed condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: Metformin SR 750mg; Drug: Rosuvastatin 10mg

INTERVENTIONS:
Drug: HCP1201 750/10mg — 750mg Metformin/10mg rosuvastatin fixed dose combination tablet orally in the morning on day1 or day8.
  Arms: HCP1201
Drug: Metformin SR 750mg — Co-administration of Metformin 750mg and Rosuvastatin 10mg orally in the morning on day1 or day8.
  Other Names: Glucophage SR 750 mg
  Arms: Metformin and Rosuvastatin
Drug: Rosuvastatin 10mg — Co-administration of Metformin 750mg and Rosuvastatin 10mg orally in the morning on day1 or day8.
  Other Names: Crestor 10mg
  Arms: Metformin and Rosuvastatin

SUMMARY:
To compare the pharmacokinetic characteristics between HCP1201 tablet 750/10 mg and co-administration of metformin 750 mg plus rosuvastatin 10 mg under fed state condition.

DETAILED DESCRIPTION:
An Open-label, Randomized, Single-dose Crossover Study to Compare the Pharmacokinetics After the Administration of HCP1201 Tablet 750/10 mg and Coadministration of Metformin SR 750 mg and Rosuvastatin 10 mg in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer, age 20~55 years
* The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 27 kg/m2
* Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial.

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study
* History of relevant drug allergies or clinically significant hypersensitivity reaction.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
metformin, rosuvastatin Cmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
metformin, rosuvastatin AUClast | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h

SECONDARY OUTCOMES:
Metformin, rosuvastatin Tmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin T1/2 | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin AUCinf | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Ryul Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea